CLINICAL TRIAL: NCT00179400
Title: The Role of Acute Combined Peroxisome Proliferator-Activated Receptors (PPAR) Alpha and Gamma Stimulation on Insulin Action in Humans
Brief Title: The Role of Acute Combined PPAR Alpha and Gamma Stimulation on Insulin Action in Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Meredith Hawkins, Professor of Medicine, Albert Einstein College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2000-200
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; 2,4-thiazolidinedione; Glucose Clamp Technique

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pioglitazone (Active Comparator): Participants received Pioglitazone 45 mg via oral capsule daily for 10 or 21 days in randomized, placebo-controlled crossover fashion, separated by a wash-out period.
  The investigators used a research procedure called a "pancreatic clamp" study to study the effects of the pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone produced in the pancreas that regulates the amount of glucose in the blood) were infused with an intravenous catheter, and blood samples were collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are related to glucose metabolism.
  Interventions: Drug: Pioglitazone; Procedure: Pancreatic Clamp Study
- Placebo (Placebo Comparator): Participants received matched placebo via oral capsule daily for 10 or 21 days in randomized, placebo-controlled crossover fashion, separated by a wash-out period.
  The investigators used a research procedure called a "pancreatic clamp" study to study the effects of the pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone produced in the pancreas that regulates the amount of glucose in the blood) were infused with an intravenous catheter, and blood samples were collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are related to glucose metabolism.
  Interventions: Drug: Placebo; Procedure: Pancreatic Clamp Study

INTERVENTIONS:
Drug: Pioglitazone — This was a randomized placebo-controlled crossover study in which subjects received both agents in random order, separated by a wash-out period. Following 10 or 21 days' intervention, subjects underwent a pancreatic clamp study.
  Other Names: Actos, Thiazolidinedione
  Arms: Pioglitazone
Drug: Placebo — This was a randomized placebo-controlled crossover study in which subjects received both agents in random order, separated by a wash-out period. Following 10 or 21 days' intervention, subjects underwent a pancreatic clamp study.
  Other Names: Control
  Arms: Placebo
Procedure: Pancreatic Clamp Study — During the clamp procedure, glucose (a sugar) and insulin were infused with an IV catheter, and blood samples were collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
  Other Names: Glucose clamp technique

SUMMARY:
The purpose of this study is to investigate the acute effects of the thiazolidinedione agent pioglitazone (which has combined PPAR alpha and gamma stimulation) on insulin's ability to suppress glucose production, stimulated glucose uptake, and impact a number of other metabolically important endpoints, including production of adiponectin (a protein hormone which regulates sugar levels and fatty acid breakdown) in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
Participants in this study were given a supply of either pioglitazone (a medication used to treat diabetes) or matched placebo for a duration of 10 days or 21 days. Changes to the body's response to insulin in the liver and in peripheral tissues (eg, muscle and fat) will be measured using a procedure called a pancreatic clamp. During the clamp procedure, glucose (a sugar) and insulin were infused with an intravenous catheter, and blood samples were collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism. Small amounts of muscle and fat tissue were also taken during this study to measure changes in gene expression after taking the medication/placebo.

ELIGIBILITY:
Inclusion Criteria:

• Individuals with Type 2 Diabetes

Exclusion Criteria:

* Individuals with bleeding disorders including gastrointestinal reflux disease (GERD), peptic ulcer disease (PUD), any gastrointestinal (GI) bleeding
* High blood pressure
* History of Coronary Artery Disease or chest pain on exertion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-12 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Hawkins, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 26 adult volunteers with type 2 diabetes completed the 10-day and/or the 21-day protocols. 13 participants completed the 10-day studies, and 13 completed the 21-day studies. Three subjects participated in both the 10-day and 21-day studies, more than six months apart.
Groups:
- 2000-200 10-day Study Only; 2000-200 10-day and 21-day Study: Participants received either 45mg of Pioglitazone (pio) or Placebo (matched to Pioglitazone) via oral capsule daily for 10 days, in randomized, placebo-controlled, cross-over fashion. Following a 4 week wash-out period, participants were crossed over to the corresponding intervention (45mg of Pioglitazone or Placebo) via oral capsule daily for 10 days.
  The investigators used a research procedure called a "pancreatic clamp" study to investigate the effects of pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
- 2000-200 21-day Study Only: Participants received either 45mg of Pioglitazone (pio) or Placebo (matched to Pioglitazone) via oral capsule daily for 21 days, in randomized, placebo-controlled, cross-over fashion. Following a 4 week wash-out period, participants were crossed over to the corresponding intervention (45mg of Pioglitazone or Placebo) via oral capsule daily for 21 days.
  The investigators used a research procedure called a "pancreatic clamp" study to study the effects of pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
Period: Overall Study
Arm/Group | 2000-200 10-day Study Only | 2000-200 21-day Study Only | 2000-200 10-day and 21-day Study
Started (3 participants from the 2000-200 10-day only study arm/group were enrolled into the 2000-200 21-day only study arm/group following a washout period of >6 months.) | 13 | 13 | 0
Placebo First 10 Day | 6 | 0 | 0
Pioglitazone First 10 Day | 7 | 0 | 0
Placebo First 21 Day | 0 | 6 | 1
Pioglitazone First 21 Day | 0 | 7 | 2
Completed | 13 | 13 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 26 adult participants with type 2 diabetes were enrolled in the 10-day and/or the 21-day studies, with a wash-out period of at least 4 weeks between Pioglitazone and Placebo. Three participants in the 10-day study also participated in the 21-day study following a washout period of > 6 months.
Groups:
- 2000-200 10-day Study: Participants received either 45mg of Pioglitazone (pio) or Placebo (matched to Pioglitazone) via oral capsule daily for 10 days, in randomized, placebo-controlled, cross-over fashion. Following a 4 week wash-out period, participants were crossed over to the corresponding intervention (45mg of Pioglitazone or Placebo) via oral capsule daily for 10 days.
  The investigators used a research procedure called a "pancreatic clamp" study to investigate the effects of pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
- 2000-200 21-day Study: Participants received either 45mg of Pioglitazone (pio) or Placebo (matched to Pioglitazone) via oral capsule daily for 21 days, in randomized, placebo-controlled, cross-over fashion. Following a 4 week wash-out period, participants were crossed over to the corresponding intervention (45mg of Pioglitazone or Placebo) via oral capsule daily for 21 days.
  The investigators used a research procedure called a "pancreatic clamp" study to investigate the effects of pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
- Total: Total of all reporting groups
Arm/Group | 2000-200 10-day Study | 2000-200 21-day Study | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Full Range); unit: years] — A total of 26 adult participants with type 2 diabetes were enrolled in the 10-day and/or the 21-day studies, with a wash-out period of at least 4 weeks between Pioglitazone and Placebo. Three participants in the 10-day study also participated in the 21-day study following a washout period of > 6 months. Population: For age, the mean and measure of dispersion were reported for the 16 participants completing the 21-day study of pioglitazone/placebo. For the 13 participants completing the 10-day study of pioglitazone/placebo, the mean age and standard error were also reported.
  years | 45.85 [45 to 50] | 47.88 [45 to 50] | 46.86 [45 to 50]
Sex: Female, Male [Count of Participants; unit: Participants] — A total of 26 adult participants with type 2 diabetes were enrolled in the 10- and/or the 21-day studies. Three of the 26 participated in both the 21- and 10- day studies, with a wash-out period of > 6 months between studies. Population: For baseline sex/gender, the number is reported for the 13 participants completing the 21-day course, for the 10 participants completing the 10-day course, and 3 participants completing both 10- and 21-day course of pioglitazone/placebo intervention. Total number of participants is 26.
  Participants
    Female | 8 | 8 | 16
    Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: number of participants] — A total of 26 adult participants with type 2 diabetes were enrolled in the 10-day and/or the 21-day studies, with a wash-out period of at least 4 weeks between Pioglitazone and Placebo. Three participants in the 10-day study also participated in the 21-day study following a washout period of > 6 months.
  number of participants
    United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Endogenous Glucose Production (EGP)
Description: EGP (a measure of the body's production of sugar) was measured by using a 6-hour stepped pancreatic clamp procedure under various treatment conditions (e.g., Pioglitazone or placebo at 10-days and/or 21-days), by monitoring the level of a non-radioactive, naturally occurring form of glucose (sugar). The relevant data at the end of each last 60 minute bin of each run was reported for each of the four groups up to 6 hours. Results are summarized by study arm/group and reported in milligrams/kilograms/minute (mg/kg/min).
Time Frame: Up to 6 hours
Measure: Mean (Standard Error); unit: mg/kg/min
Groups:
- 2000-200 Study 10-day Pioglitazone: Participants received Pioglitazone (pio) 45mg via oral unmarked capsule daily for 10 days with a wash-out period of at least 4 weeks between studies. This is a randomized, double blinded, cross-over study, so subjects who participated in the pioglitazone intervention also participated in the placebo intervention. Either placebo or pioglitazone was administered to each subject randomly for the study.
  The investigators used a research procedure called a "pancreatic clamp" study to study the effects of pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
- 2000-200 Study 10-day Placebo: Participants received placebo via oral unmarked capsule daily for 10 days with a wash-out period of at least 4 weeks between studies. This is a randomized, double blinded, cross-over study, so subjects who participated in the pioglitazone intervention also participated in the placebo intervention. Either placebo or pioglitazone was administered to each subject randomly for the study.
  The investigators used a research procedure called a "pancreatic clamp" study to study the effects of pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
- 2000-200 Study 21-day Pioglitazone: Participants received Pioglitazone (pio) 45mg via oral unmarked capsule daily for 21 days with a wash-out period of at least 4 weeks between studies. This is a randomized, double blinded, cross-over study, so subjects who participated in the pioglitazone intervention also participated in the placebo intervention. Either placebo or pioglitazone was administered to each subject randomly for the study.
  The investigators used a research procedure called a "pancreatic clamp" study to study the effects of pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
- 2000-200 Study 21-day Placebo: Participants received placebo via oral unmarked capsule daily for 21 days with a wash-out period of at least 4 weeks between studies. This is a randomized, double blinded, cross-over study, so subjects who participated in the pioglitazone intervention also participated in the placebo intervention. Either placebo or pioglitazone was administered to each subject randomly for the study.
  The investigators used a research procedure called a "pancreatic clamp" study to study the effects of pioglitazone. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
Arm/Group | 2000-200 Study 10-day Pioglitazone | 2000-200 Study 10-day Placebo | 2000-200 Study 21-day Pioglitazone | 2000-200 Study 21-day Placebo
Number analyzed (Participants) | 13 | 13 | 16 | 16
mg/kg/min | 1.26 (0.19) | 1.25 (0.20) | 0.90 (0.13) | 1.48 (0.18)

2. Primary Outcome: Glucose Rates of Disappearance (Rd)
Description: Glucose rates of disappearance were measured using a stepped pancreatic clamp study procedure under various treatment conditions (e.g., Pioglitazone or placebo at 10-days and/or 21-days) by monitoring the level of a non-radioactive, naturally occurring form of glucose (sugar). For purposes of this study, the most relevant data for the final hour is summarized within each study Pioglitazone and Placebo study arm/group, respectively. Results are summarized by study arm/group and reported in milligrams/kilograms/minute (mg/kg/min).
Time Frame: Up to 6 hours
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | 2000-200 Study 10-day Pioglitazone | 2000-200 Study 10-day Placebo | 2000-200 Study 21-day Pioglitazone | 2000-200 Study 21-day Placebo
Number analyzed (Participants) | 13 | 13 | 16 | 16
mg/kg/min | 3.9 (0.15) | 3.6 (0.10) | 3.90 (0.15) | 3.60 (0.10)

3. Secondary Outcome: Gene Expression in Both Whole Fat Tissue and Isolated Macrophages
Description: Gene expression of inflammatory markers in both whole fat tissue and isolated macrophages were studied by quantitative, real-time reverse transcriptase polymerase chain reaction (RT-PCR) in placebo and Pioglitazone groups of either 10- or 21-day study. The reporting data was calculated as the ratio between the target genes and housekeeping genes in either the 10- or 21-day study.
Time Frame: Outcome was compared prior to and post 10-day or 21-day administration of either placebo or Pioglitazone
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | 2000-200 Study 10-day Pioglitazone | 2000-200 Study 10-day Placebo | 2000-200 Study 21-day Pioglitazone | 2000-200 Study 21-day Placebo
Number analyzed (Participants) | 13 | 13 | 16 | 16
ratio
  Adipose tissue macrophage MCP-1 | 0.80 (0.60) | 1.90 (0.50) | 0.07 (0.01) | 0.11 (0.02)
  Adipose tissue macrophage CCR2 | 0.009 (0.001) | 0.023 (0.007) | 0.0020 (0.0005) | 0.0040 (0.0005)
  Adipose tissue hyaluronan synthase expression | 0.007 (0.001) | 0.015 (0.002) | 0.013 (0.007) | 0.019 (0.006)
  Adipose tissue hyaluronan receptor CD44 expression | 0.150 (0.075) | 0.225 (0.025) | 0.050 (0.01) | 0.10 (0.01)
  Macrophage CD14 expression | 0.79 (0.01) | 0.84 (0.02) | 0.07 (0.01) | 0.11 (0.02)
  Macrophage CD68 expression | 0.23 (0.07) | 0.26 (0.02) | 0.20 (0.05) | 0.40 (0.1)
  Whole adipose tissue DEC205 | 0.0009 (0.0002) | 0.0016 (0.02) | 0.0015 (0.0004) | 0.0024 (0.0003)
  Whole adipose tissue DC SIGN | 0.0007 (0.0002) | 0.001 (0.0001) | 0.005 (0.0020) | 0.0125 (0.0040)
  Whole adipose tissue MPO-3 | 0.018 (0.009) | 0.031 (0.012) | 0.009 (0.002) | 0.02 (0.004)
  Whole adipose tissue FOXP3 | 0.0005 (0.0001) | 0.0006 (0.0001) | 0.0035 (0.0010) | 0.0045 (0.0013)
  Whole adipose tissue CD25 | 0.89 (0.04) | 0.90 (0.05) | 0.0035 (0.0008) | 0.0045 (0.0013)

4. Secondary Outcome: Effects of Pioglitazone on Adipose Tissue Percentage of Macrophage Content
Description: Adipose tissue biopsy was performed on day one or on the last day (10th or 21st day) for the corresponding Pioglitazone and placebo interventions. Macrophages were stained with immunofluorescence antibody after isolation from adipose tissue and processed. The percentage of macrophage content in stromal vascular fraction cells (SVF) analyzed by Fluorescence-activated cell sorter analysis (FACS) was determined. Results are summarized by study arm/group and reported in milligrams/kilograms/minute (mg/kg/min).
Time Frame: Assessed at day 1 prior to the intervention and on day 10 or 21 following the intervention, day 10 or 21 following the intervention reported
Population: Day 1 macrophage data was not collected and reported.
Measure: Mean (Standard Error); unit: percentage of macrophage content
Arm/Group | 2000-200 Study 10-day Pioglitazone | 2000-200 Study 10-day Placebo | 2000-200 Study 21-day Pioglitazone | 2000-200 Study 21-day Placebo
Number analyzed (Participants) | 13 | 13 | 16 | 16
percentage of macrophage content | 10.20 (1.6) | 12.00 (1.9) | 4.20 (2.80) | 13.50 (1.50)

5. Secondary Outcome: Adipose Tissue Percentage of Macrophage Content
Description: Adipose tissue percentage of macrophage content was analyzed by Immuno-fluorescence staining (iNOS+ and CD68+). Both the immuno-fluorescence stained macrophages and all other stained cells will be counted after staining. The percentage of macrophage content will be calculated as the the ratio between the number of macrophage and all other cells.
Time Frame: Outcome was compared between Pioglitazone and placebo group prior to and after 21-day administration
Population: Due to the unsuccessful IHF assay macrophage % content data was not collected for the 10-day study.
Measure: Mean (Standard Error); unit: percentage of macrophage content
Arm/Group | 2000-200 Study 21-day Pioglitazone | 2000-200 Study 21-day Placebo
Number analyzed (Participants) | 16 | 16
percentage of macrophage content | 18 (7) | 43 (15)

6. Secondary Outcome: Adipose Tissue Regulatory T Lymphocyte Content
Description: Adipose tissue T lymphocyte content (%) was analyzed by Immunohistochemistry (IHC) staining with Treg-specific marker FOXP3
  Both the IHC FOXP3 stained T lymphocyte and all other stained cells will be counted after staining. The percentage of T lymphocyte content will be calculated as the the ratio between the number of T lymphocyte and all other cells.
Time Frame: Outcome was compared between Pioglitazone and placebo group prior to and after 21-day administration
Population: Due to the unsuccessful IHC assay, T lymphocyte % content was unable to be collected for the 10-day study.
Measure: Mean (Standard Error); unit: percentage of T lymphocyte content
Arm/Group | 2000-200 Study 21-day Pioglitazone | 2000-200 Study 21-day Placebo
Number analyzed (Participants) | 16 | 16
percentage of T lymphocyte content | 14 (3) | 17 (5)

ADVERSE EVENTS:
Time Frame: Up to 10 days for participants in 10-day treatment and 21 days for participants in 21-day treatment.
Arm/Group | 2000-200 Study 10-day Pioglitazone | 2000-200 Study 10-day Placebo | 2000-200 Study 21-day Pioglitazone | 2000-200 Study 21-day Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/16 | 1/16
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2000-200 Study 10-day Pioglitazone (N=13) | 2000-200 Study 10-day Placebo (N=13) | 2000-200 Study 21-day Pioglitazone (N=16) | 2000-200 Study 21-day Placebo (N=16)
Hypotensive Episode (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Following clamp study, Blood Pressure (BP) 64/40, Heart Rate (HR) 88. Subject had no intake of oral fluids since 11p the night before study. Following infusion of 3 liters of intravenous fluid, subject was discharged in stable condition. BP 110/68.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No